CLINICAL TRIAL: NCT06358807
Title: Clinical Efficacy of Arthroscopic Microfracture Combined With Local Injection of Platelet Rich Plasma Gel in Treatment of Osteochondral Lesion of the Talus: A Randomized Control Trial
Brief Title: Microfracture With Platelet Rich Plasma Gel Injection for Osteochondral Lesion of the Talus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M2023438
Record Dates: First submitted 2024-04-07; First posted 2024-04-11 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-03

CONDITIONS: Osteochondral Lesion of Talus; Microfractures; Platelet Rich Plasma
Keywords: Osteochondral Lesion of Talus; Microfractures; Platelet Rich Plasma; Arthroscopic Techniques; Clinical Efficacy
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microfracture with PRP (Experimental): Arthroscopic microfracture:
  An anteromedial portal and an anterolateral portal are routinely established. A diagnostic arthroscopy is performed. Defects of superficial cartilage, cystic components, and necrotic bone are debrided arthroscopically with curette and shaver to a stable circumferential rim. Microfracture awls are introduced and subchondral channels to 4-6 mm in depth are created, spacing the channels 3 to 5 mm apart across the entire surface of the lesion.
  PRP preparation and local injection:
  PRP is harvested using a PRP preparation kit via centrifugation. Fifty milliliters of autologous venous blood are drawn from the patient and processed. Platelet count is measured for quality control. On average 4 ml of (range 3-6) PRP is obtained and mixed with thrombin calcium agent in preparation for PRP gel. PRP gel is administered to the injured area using a blunt and long-tip injector, with direct visualization under arthroscope.
  Interventions: Procedure: Arthroscopic microfracture with intraoperative local PRP gel injection
- Isolated microfracture (Active Comparator): Arthroscopic microfracture:
  An anteromedial portal and an anterolateral portal are routinely established. A diagnostic arthroscopy is performed. Defects of superficial cartilage, cystic components, and necrotic bone are debrided arthroscopically with curette and shaver to a stable circumferential rim. Microfracture awls are introduced and subchondral channels to 4-6 mm in depth are created, spacing the channels 3 to 5 mm apart across the entire surface of the lesion.
  Interventions: Procedure: Isolated microfracture

INTERVENTIONS:
Procedure: Arthroscopic microfracture with intraoperative local PRP gel injection — Arthroscopic microfracture:
  An anteromedial portal and an anterolateral portal are routinely established. A diagnostic arthroscopy is performed. Defects of superficial cartilage, cystic components, and necrotic bone are debrided arthroscopically with curette and shaver to a stable circumferential rim. Microfracture awls are introduced and subchondral channels to 4-6 mm in depth are created, spacing the channels 3 to 5 mm apart across the entire surface of the lesion.
  PRP preparation and local injection:
  PRP is harvested using a PRP preparation kit via centrifugation. Fifty milliliters of autologous venous blood are drawn from the patient and processed. Platelet count is measured for quality control. On average 4 ml of (range 3-6) PRP is obtained and mixed with thrombin calcium agent in preparation for PRP gel. PRP gel is administered to the injured area using a blunt and long-tip injector, with direct visualization under arthroscope.
  Arms: Microfracture with PRP
Procedure: Isolated microfracture — Arthroscopic microfracture:
  An anteromedial portal and an anterolateral portal are routinely established. A diagnostic arthroscopy is performed. Defects of superficial cartilage, cystic components, and necrotic bone are debrided arthroscopically with curette and shaver to a stable circumferential rim. Microfracture awls are introduced and subchondral channels to 4-6 mm in depth are created, spacing the channels 3 to 5 mm apart across the entire surface of the lesion.
  Arms: Isolated microfracture

SUMMARY:
The goal of this clinical trial is to learn if combined local injection of platelet rich plasma (PRP) gel adds clinical efficacy to isolated arthroscopic microfracture in treatment of osteochondral lesion of the talus (OLT). The interface integration of the injured area will also be assessed via radiographic follow-up. The main questions it aims to answer are:

* Does arthroscopic microfracture combined with PRP gel injection improve ankle function of participants based on American Orthopedic Foot and Ankle Society (AOFAS) Score?
* Does arthroscopic microfracture combined with PRP gel injection improve interface integration of the injured cartilage on magnetic resonance imaging (MRI)? Researchers will compare arthroscopic microfracture with concomitant local injection of PRP gel to isolated microfracture to see if intraoperative PRP gel injection adds clinical efficacy to isolated arthroscopic microfracture in treatment of OLT.

Participants will:

* Undergo either isolated arthroscopic microfracture or microfracture with intraoperative injection of PRP gel
* Receive clinical follow-up 3, 6, 12, and 24 months after surgery and answer scales of ankle function assessment
* Take MRI preoperatively and 6, 12 and 24 months after surgery

ELIGIBILITY:
Inclusion Criteria:

* Chronic ankle pain, diagnosed as osteochondral lesion of the talus;
* Lesion size ≤ 1.5 cm2 or the diameter of the lesion ≤ 1.5 cm;
* Conservative treatment of at least 3 months fails to relieve symptoms;
* Willingness to voluntarily participate in the trial and to sign informed consent.

Exclusion Criteria:

* Varus or valgus deformity of the ankle of more than 5 degrees;
* Grade III injury of the lateral collateral ligament of ankle;
* Chronic synovitis (rheumatoid arthritis, pigmented villous nodular synovitis, etc.);
* Joint fibrosis, stiffness, and significantly restricted range of motion;
* Evidence of moderate to severe knee osteoarthritis on plain radiographs;
* Failure to complete the rehabilitation protocol as required;
* Patient medically not fit for surgery, radiographs or MRI;
* For women, pregnant, planning to be pregnant or lactating.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
American Orthopedic Foot and Ankle Society Score (AOFAS) | Pre-surgery and 3, 6, 12 and 24 months after surgery
  The scale of AOFAS score will be answered by participants during clinic follow-up preoperatively, and 3, 6, 12 and 24 months after surgery. The primary outcome measure will be the AOFAS collected 24 months post-surgery.

SECONDARY OUTCOMES:
Foot and Ankle Outcome Score (FAOS) | Pre-surgery and 3, 6, 12 and 24 months after surgery
  The scale of FAOS score will be answered by participants during clinic follow-up preoperatively, and 3, 6, 12 and 24 months after surgery.
Ankle Activity Score (AAS) | Pre-surgery and 3, 6, 12 and 24 months after surgery
  The scale of AAS score will be answered by participants during clinic follow-up preoperatively, and 3, 6, 12 and 24 months after surgery.
Visual Analogue Scale (VAS) | Pre-surgery and 3, 6, 12 and 24 months after surgery
  The scale of VAS score will be answered by participants during clinic follow-up preoperatively, and 3, 6, 12 and 24 months after surgery.
Patient Satisfaction | Final follow-up (24 months after surgery)
  Patient satisfaction will be graded as 0-10 and collected 24 months after surgery.
Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) | Twelve and 24 months after surgery
  MOCART score will be assessed on magnetic resonance imaging 12 and 24 months after surgery.
Return-to-Sport Rate | Final follow-up (24 months after surgery)
  The rate and time point of participants returning to sports will be continuously followed during clinic follow-up and will be overall collected 24 months after surgery.
Complications | Final follow-up (24 months after surgery)
  Complications, including infection,hematoma, stiffness, recurrent ankle pain will be continuously followed during clinic follow-up and will be overall collected 24 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Qinwei Guo, MD, Principal Investigator — Department of Sports Medicine, Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China